CLINICAL TRIAL: NCT06242457
Title: Poorly Differentiated Adenocarcinoma of the Jejunum in a Patient With Peutz-Jeghers Syndrome: A Case Report
Status: Completed | Type: Observational
Sponsor: Haramaya Unversity (Other)
Responsible Party: Principal Investigator, Fufa Miresa, Principal investigator, Assistant professor of general surgery, Haramaya Unversity
Other Study IDs: HU
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Peutz-Jeghers Syndrome
MeSH Terms: conditions — Peutz-Jeghers Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study is a case report of one of the rarest risk factor, Peutz-Jeghers syndrome, of small bowel malignancy detected in a patient with poorly differentiated adenocarcinoma of small bowel(jejunum)

DETAILED DESCRIPTION:
Case presentation: A 25-year-old male patient presented to the emergency department with generalized peritonitis caused by a perforated jejunal mass. The patient underwent an emergency exploratory laparotomy. There was 800 ml of thin pus in the peritoneal cavity and 5 cm by 6 cm perforated mass over the jejunum, 30cm from the ligament of the treitz, which extends to the mesentery. Palpable jejunal mesenteric lymphadenopathies were found. There were palpable intraluminal polyps with an inverted serosal surface for some of them, which were identified as 10cm proximal and 20cm distal to the mass. The pus was sucked out, and the mass was resected with its mesenteric lymph nodes and segments containing polyps, a total of 40cm of jejunum. Subsequently, end-to-end hand-sewn anastomosis was performed, and the abdomen was closed. The histopathology report showed poorly differentiated adenocarcinoma, stage IIIC (PT3, PN2), and Peutz-Jeghers polyps, suggesting Peutz-Jeghers syndrome. Lympho-vascular invasion was also noted. The tumor has affected seven of the 12 lymph nodes that have been identified. After 6weeks of uneventful follow-up at the surgical referral clinic, the patient was referred to the oncology department for adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* not necessary

Exclusion Criteria:

* not necessary

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: New patient came to emergency department as routine activity.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Complete resection of adenocarcinomas located in the jejunum or ileum is associated with 5-year survival rates of 20% to 30%. | 5months
  Even though small bowel malignancy is a rare entity, early detection is a challenging issue, especially when it happens below the ligaments of the trietz. Peutz-Jeghers syndrome was a potential risk factor in our case.

CONTACTS AND LOCATIONS:
Locations (1):
- Haramaya University, Harar, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: after publication